CLINICAL TRIAL: NCT06544486
Title: Clinical Evaluation of Contemporary Ion Releasing Restorative Materials in Primary Molars Subjected to Selective Caries Removal: A Randomized Clinical Trial
Brief Title: Contemporary Restorative Materials in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Zulfikar Zahit Ciftci, Head of Pediatric Dentistry, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDH- 2022-5832
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries
Keywords: Cention N; Resin-modified glass-ionomer cement; Hybrid glass-ionomer cement; Zinc reinforced glass-ionomer cement; Primary Molar Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Masking Description: The materials were visually different from each other, which allowed the investigators to identify each material. As a result, masking could only be performed with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Device: Hybrid Glass-ionomer Cement (Equia Forte HT) (Experimental): The material in capsule form was placed in the mixer (Ultramat 2, SDI, Australia) and mixed for 10 seconds, and applied to the cavity in a single step. The restorative material was polymerized for 20 seconds using an LED light device (VALO, Ultradent, Utah, USA). Equia Forte Coat was applied and polymerized for 20 seconds.
  Interventions: Procedure: Caries Removal; Procedure: Filling
- Device: Resin-Modified Glass-ionomer Cement (Fuji II LC) (Experimental): The material in capsule form was mixed in the mixer (Ultramat 2, SDI, Australia) for 10 seconds, and applied to the cavity in a single step. Polymerization was achieved using an LED light device (VALO, Ultradent, Utah, USA) for 20 seconds.
  Interventions: Procedure: Caries Removal; Procedure: Filling
- Device: Bioactive Glass-Containing Alkasite (Cention N) (Experimental): The material was mixed using a plastic spatula on a mixing pad or glass with a powder-to-liquid ratio of 1:1 until it reached a homogeneous consistency, which took approximately 45 -60 seconds. Then the material was applied to the cavity and allowed to set for its self-curing time of 4 and a half minutes.
  Interventions: Procedure: Caries Removal; Procedure: Filling
- Device: Zinc-Reinforced High-Viscosity Glass-ionomer Cement (ChemFil Rock) (Experimental): The material in capsule form was placed in the mixer (Ultramat 2, SDI, Australia) and mixed for 12 seconds, and applied to the cavity in a single step. In addition to the 90-second working time, an additional 4 and a half minutes were allowed for the material to cure.
  Interventions: Procedure: Caries Removal; Procedure: Filling

INTERVENTIONS:
Procedure: Caries Removal — The cavity preparation and restoration were performed by a single operator. Infected dentin tissue was selectively removed. The differentiation between infected and affected dentin was determined by the clinician through the visual-tactile method.Isolation was achieved with cotton rolls and suction.
Procedure: Filling — Sectional matrix systems and interdental wedges were used to achieve an anatomical contour and contact. Then, the selected materials were placed in the cavity according to the manufacturers' recommendations.

SUMMARY:
This randomized controlled trial aims to compare the clinical effectiveness of four ion-releasing restorative materials in the proximal cavities of primary molars that underwent selective caries removal. The main questions to answer are:

* Will there be any difference among the restorative materials clinical succes in the means of modified United States Public Health Services (USPHS) criteria for dental restorations?
* Will there be any difference among the restorative materials in the means of preservation of pulpal vitality? Eighty six children (262 teeth), between 5 and 9 years old (7.15±1.14) enrolled for the study. Researchers will compare the clinical performance of restorative materials, (1:Equia Forte HT; 2: Fuji II LC; 3: Cention N; 4: ChemFil Rock), applied to the proximal cavities of primary molars following selective caries removal, according to the modified USPHS criteria.

Participants will:

- visit the clinic 1st,3rd,6th,12th,18th,24th,30th and 36th months after the restoration.

ELIGIBILITY:
Inclusion Criteria:

For participants:

* no known or suspected history of allergy to medications or restorative materials
* no habits of teeth grinding or clenching
* presence of at least one interproximal carious lesion

For teeth:

* carious lesion reaching at least 1/2 dentin
* in contact with adjacent teeth and in occlusion with antagonist teeth
* have no pathological mobility
* periodontally healthy
* no symptoms of pulpal pathology
* physiological root resorption should not exceed one-third of the root length if seen
* permanent tooth germ present below the tooth

Exclusion Criteria:

* did not attend their follow-up appointments

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of the filling materials according to the modified USPHS criteria | Evaluations were conducted at the 1st, 3rd, 6th, 12th, 18th, 24th, 30th and 36th months.
  Restorations were evaluated for retention, marginal discoloration, marginal adaptation, color stability, secondary caries, and postoperative sensitivity according to the modified USPHS with scores assigned as follows: the best being Alpha and the worst being Charlie. Each restoration received a score of Alpha, Bravo, or Charlie at each time interval.

SECONDARY OUTCOMES:
Preservation of pulpal vitality | Evaluations were conducted at the 1st, 3rd, 6th, 12th, 18th, 24th, 30th and 36th months.
  The modified USPHS criteria do not include the measure of pulpal vitality when evaluating the success of restorations. However, maintaining pulpal vitality is also a criterion for the success of a restoration and is assessed not by a graded score but by the presence or absence of symptoms and findings. In this study, pulpal vitality was clinically evaluated based on the presence or absence of percussion sensitivity, palpation sensitivity, gingival redness, fistula or abscess. If percussion sensitivity, palpation sensitivity, or the formation of a fistula or abscess were present, the restoration was classified as unsuccessful regarding pulpal vitality. In cases of gingival redness or unclear clinical symptoms, a periapical radiograph was taken. If presence or absence of radiolucency in the periapical or furcal area was detected in the radiograph, the restoration was classified as unsuccessful regarding pulpal vitality.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfikar Zahit Ciftci, Phd, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)